CLINICAL TRIAL: NCT05059600
Title: Assessment of Safe-use Conditions for Administration of ZULRESSO in a Home Setting
Brief Title: A Study To Assess The Safe-Use Conditions For Administration of ZULRESSO® in a Home Setting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 547-PPD-404
Record Dates: First submitted 2021-09-17; First posted 2021-09-28 (Actual); Results first posted 2023-07-19 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2023-06

CONDITIONS: Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum | interventions — brexanolone; Pregnanolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ZULRESSO® (Experimental): Participants received a 60-hour single continuous intravenous (IV) infusion of ZULRESSO®, at 30 micrograms per kilogram per hour (mcg/kg/hour) (0 to 4 hours), at 60 mcg/kg/hour (4 to 24 hours), at 90 mcg/kg/hour (24 to 52 hours), followed by a dose taper to 60 mcg/kg/hour (52 to 56 hours), and 30 mcg/kg/hour (56 to 60 hours) during the study.
  Interventions: Drug: ZULRESSO®

INTERVENTIONS:
Drug: ZULRESSO® — Intravenous infusion of ZULRESSO®.
  Other Names: Allopregnanolone; Brexanolone; SAGE-547

SUMMARY:
The primary purpose of this study was to evaluate whether the safe-use conditions for administration of brexanolone (ZULRESSO®) can be implemented in a home setting.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory female ≥18 years of age.
2. Participant has a current diagnosis of postpartum depression (PPD), as confirmed by the investigator.
3. Participant agrees not to be the primary caregiver of any dependents during the infusion and must be accompanied by another adult (other than the home healthcare provider) during interactions with their child(ren).
4. Participant has no history of sleep apnea or any clinically significant respiratory conditions.
5. Participant agrees to refrain from the use of central nervous system depressants, such as opioids, benzodiazepines, sleep aids and from drinking alcohol during the infusion.
6. Participant is suitable for administration of ZULRESSO® in a home setting, as per the judgement of the investigator.
7. Participant's home is suitable and has necessary provisions for administration of ZULRESSO® and meets the following criteria:

   * safe environment for the home infusion provider staff.
   * access to a working telephone.
   * electricity and grounded electrical outlets.
   * running water.
   * access to back-up emergency services (911 service or ambulance availability).
   * sanitary environment.
8. Participant agrees to stay at home until the end-of-study visit has been completed, except for a medical emergency.
9. Participant must have a negative pregnancy test at screening and on Day 1 prior to the start of the ZULRESSO® infusion.

Exclusion Criteria:

1. Participant has end stage renal failure.
2. Participant has known allergy to progesterone or allopregnanolone or any excipients in the brexanolone injection.
3. Participant is currently at risk of suicide, as judged by the investigator, or has attempted suicide associated with the current episode of PPD.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 52 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2022-07-14 (Actual); Study Completion 2022-07-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Sage Investigational Site, Culver City, California
  - Virtual Site (recruiting nationwide), Culver City, California
  - Sage Investigational Site, Miramar, Florida
  - Sage Investigational Site, Pompano Beach, Florida
  - Sage Investigational Site, New York, New York
  - Sage Investigational Site, League City, Texas

IPD SHARING:
Plan to Share IPD: No
Data sharing will be consistent with the results submission policy of ClinicalTrials.gov

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 5 active clinical sites in the United States from 08 October 2021 to 14 July 2022.
Pre-assignment Details: A total of 80 participants were screened, of which 52 were enrolled and 42 were treated.
Period: Overall Study
Arm/Group | ZULRESSO®
Started | 52
Treated | 42
Completed | 42
Not Completed | 10
Not completed — Enrolled but not Treated | 10

BASELINE CHARACTERISTICS:
Population: Safety Set included all participants who were administered ZULRESSO®.
Groups:
- ZULRESSO®: Participants received a 60-hour single continuous IV infusion of ZULRESSO®, at 30 mcg/kg/hour (0 to 4 hours), at 60 mcg/kg/hour (4 to 24 hours), at 90 mcg/kg/hour (24 to 52 hours), followed by a dose taper to 60 mcg/kg/hour (52 to 56 hours), and 30 mcg/kg/hour (56 to 60 hours) during the study.
Arm/Group | ZULRESSO®
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.9 (5.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 33
  Black or African American | 6
  Asian | 1
  American Indian or Alaska Native | 0
  Native Hawaiian or Other Pacific Islander | 0
  Other | 1
  Not Specified | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With At Least One Treatment-Emergent Adverse Event (TEAE) Leading to Dose Interruption/Discontinuation
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical investigation participant administered with a pharmaceutical product that does not necessarily have a causal relationship with this treatment. A TEAE was defined as an AE with onset after the start of investigational product, or any worsening of a preexisting medical condition/AE with onset after the start of investigational product and throughout the study. Percentages are rounded off to the nearest single decimal.
Time Frame: Up to Day 3
Population: Safety Set included all participants who were administered ZULRESSO®.
Measure: Number; unit: percentage of participants
Groups:
- ZULRESSO®: Participants received a 60-hour single continuous IV infusion of ZULRESSO®, at 30 mcg/kg/hour (0 to 4 hours), at 60 mcg/kg/hour (4 to 24 hours), at 90 mcg/kg/hour (24 to 52 hours), followed by a taper to 60 mcg/kg/hour (52 to 56 hours), and 30 mcg/kg/hour (56 to 60 hours) during the study.
Arm/Group | ZULRESSO®
Number analyzed (Participants) | 42
percentage of participants | 7.1

2. Secondary Outcome: Percentage of Participants With Nonadherence With the Safe-Use Conditions for Administration of ZULRESSO®
Description: Nonadherence was defined by failure of any of following:
  * Home infusion provider to train all pharmacy and home healthcare providers (HHPs) in dispensing/administration of ZULRESSO® on risk of excessive sedation/loss of consciousness
  * HHPs to counsel participants on risk of excessive sedation/loss of consciousness
  * Deliver ZULRESSO® per protocol
  * Provide preprogrammed peristaltic pump
  * HHP:assess excessive sedation every 2 hours in planned nonsleep periods, change infusion bag per protocol, at least one HHP available in participant's home for the duration of infusion
  * Fall protocol in place
  * Monitor participants with pulse oximeter
  * Stop infusion when participant is primary caregiver of dependents and/or identification of excessive sedation/loss of consciousness/hypoxic episode
  * Caution participants post-infusion against engaging in hazardous activities requiring mental alertness
  * Complete AE of special interest/Serious AE form
  * Infusion resumed after hypoxia episode
Time Frame: Up to Day 3
Population: Safety Set included all participants who were administered ZULRESSO®.
Measure: Number; unit: percentage of participants
Arm/Group | ZULRESSO®
Number analyzed (Participants) | 42
percentage of participants | 76.19

3. Secondary Outcome: Number of Use-Related Issues Related to the Home Administration of ZULRESSO®
Description: Home healthcare provider (HHP) staff completed checklists at end of each day and/or shift to document any use-related issues throughout duration of infusion. Any use-related issues determined to be critical in nature were followed up immediately and were reported adequately. Use-related issues were categorized as Critical Use Error (UE): HHP failed to complete a task or made uncorrected use error during task that could have resulted in harm, compromised medical care, incidence of nonadherence with safe use conditions for administration of ZULRESSO, or incidence of use-related issues related to home administration of ZULRESSO; Use Difficulty (UD): HHP successfully completed a task but did so while experiencing issues/operational difficulties; Close Call (CC): HHP committed error that could have led to a task failure, but self-corrected and completed task successfully. Multiple occurrences of issue throughout a single infusion was included only once in total.
Time Frame: Up to Day 3
Population: Safety Set included all participants who were administered ZULRESSO®. Overall number of units analyzed signifies total number of use related issues.
Measure: Count of Units; unit: Issues
Units Other Than Participants: Issues
Arm/Group | ZULRESSO®
Number analyzed (Participants) | 42
Number analyzed (Issues) | 75
Issues
  Critical Use Errors (UE) | 13
  Use Difficulties (UD) | 62
  Close Calls (CC) | 0

4. Secondary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An AE was any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. TEAE was defined as an AE with onset after the start of investigational product, or any worsening of a preexisting medical condition/AE with onset after the start of investigational product and throughout the study. Percentages are rounded off to nearest single decimal.
Time Frame: Up to Day 3
Population: Safety Set included all participants who were administered ZULRESSO®.
Measure: Number; unit: percentage of participants
Arm/Group | ZULRESSO®
Number analyzed (Participants) | 42
percentage of participants | 42.9

5. Secondary Outcome: Percentage of Participants With Medication Error
Description: Medication error was any preventable event that may cause or lead to inappropriate medication use or participant harm while the medication was in the control of the healthcare professional, participant, or consumer. Percentages are rounded off to the nearest single decimal.
Time Frame: At screening and during the study (Up to Day 3)
Population: Safety Set included all participants who were administered ZULRESSO®.
Measure: Number; unit: percentage of participants
Arm/Group | ZULRESSO®
Number analyzed (Participants) | 42
percentage of participants
  At Screening | 28.6
  During the Study (Up to Day 3) | 54.8

ADVERSE EVENTS:
Time Frame: Up to Day 3
Description: Safety Set included all participants who were administered ZULRESSO®.
Arm/Group | ZULRESSO®
All-Cause Mortality (participants affected / at risk) | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 15/42
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ZULRESSO® (N=42)
Fatigue (General disorders) | 5
Infusion site pain (General disorders) | 3
Headache (Nervous system disorders) | 4
Somnolence (Nervous system disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI can either be a party and subject to the same restrictions as the institution, or if not a party, the restrictions are described on the face of the contract (i.e., PI is a contractor of the institution; PI is part of a larger group of study personnel; institution has contracted with or otherwise bound all study personnel under confidentiality obligations and requirements to vest intellectual property to the institution).

DOCUMENTS (2):
  • Study Protocol (2021-06-28): https://cdn.clinicaltrials.gov/large-docs/00/NCT05059600/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-09): https://cdn.clinicaltrials.gov/large-docs/00/NCT05059600/SAP_001.pdf